CLINICAL TRIAL: NCT02598635
Title: Effects of Cholecalciferol on Osteoprotegerin Levels and Other Clinical Outcomes in Chronic Kidney Disease Patients on Peritoneal Dialysis: a Randomized Controlled Trial
Brief Title: Effects of Cholecalciferol on Osteoprotegerin Levels in Patients on Peritoneal Dialysis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Juan C Ramirez-Sandoval, MD, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1419
Record Dates: First submitted 2015-10-31; First posted 2015-11-06 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Vitamin D Deficiency; Vascular Calcification; Renal Insufficiency; End Stage Renal Failure on Dialysis
Keywords: Cholecalciferol; peritoneal dialysis; FGF23; Calcium; Phosphorus
MeSH Terms: conditions — Vitamin D Deficiency; Vascular Calcification; Renal Insufficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cholecalciferol (Experimental): A capsule of pulverized cholecalciferol 4800 U will be administered once a day for 16 weeks. At serum calcium levels > 10.5 mg/dL (2.65 mmol/l) and/or at serum phosphorus levels > 7 mg/dL (2.26 mmol/L) capsule administration will be discontinued and restarted one month after when serum calcium levels or phosphorus levels declined to < 10.6 mg/dL and/or <7.1 mg/dL respectively.
  Interventions: Drug: Cholecalciferol
- Placebo (Placebo Comparator): An oral placebo capsule matching Cholecalciferol in terms of appearance, smell and taste will be administered once a day for 16 weeks. At serum calcium levels > 10.5 mg/dL (2.65 mmol/l) and/or at serum phosphorus levels > 7 mg/dL (2.26 mmol/L) capsule administration will be discontinued and restarted one month after when serum calcium levels or phosphorus levels declined to < 10.6 mg/dL and/or <7.1 mg/dL respectively.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cholecalciferol — Patients on peritoneal dialysis and 25-(OH) levels <20 ng/mL will received one capsule of cholecalciferol (4800 U) once a day for 16 weeks.
  Other Names: "Valmetrol-3"
  Arms: Cholecalciferol
Drug: Placebo — An oral placebo capsule matching Cholecalciferol in terms of appearance, smell and taste will be administered once a day for 16 weeks.
  Other Names: (Capsule similar to Cholecalciferol)
  Arms: Placebo

SUMMARY:
Aim: To investigate whether cholecalciferol (4800 U/daily) or placebo for 16 weeks reduces proteins levels associated with vascular calcification (osteoprotegerin, osteopontin, osteocalcin) in patients treated with peritoneal dialysis and 25(OH) vitamin D deficiency.

DETAILED DESCRIPTION:
Patients with chronic kidney disease on peritoneal dialysis have very low 25-(OH) vitamin D levels. Vitamin D deficiency may be involved in generalized atherosclerosis, vascular calcification and cardiovascular mortality. Among others, Osteoprotegerin (OPG) has been implicated in the pathogenesis leading up vessel calcification in this patients. Furthermore, very low levels of 25-(OH) vitamin D in peritoneal dialysis patients are associated with increased levels of OPG and high values of vascular calcification scores in x-rays.

It is unknown whether cholecalciferol supplementation in patients on peritoneal dialysis with low levels of 25-(OH) vitamin D could change the proteins associated with vascular calcification.

The objective is to conduct a randomized, double-blind, placebo-controlled study focusing on the impact of Cholecalciferol substitution in 25-OH vitamin D deficient peritoneal dialysis patients on circulating OPG and other osteogenic biomarkers levels during 16 weeks of intervention.

Moreover, the impact of cholecalciferol on serum calcium and phosphorus levels, Kidney Disease Quality of Life Short Form, and ultrasound characteristics of carotid arterial will be performed during the first four weeks after inclusion, and after 28 weeks postintervention.

Peritoneal dialysis patients found to have 25-(OH) vitamin D levels <20 ng/ml will be included and will be randomized to receive either oral cholecalciferol therapy or placebo. Cholecalciferol will be administered at a daily dose of 4800 IU over a time period of 16 weeks.

All in all, 58 subjects will be included in this study.

ELIGIBILITY:
Inclusion Criteria:

* Peritoneal dialysis treatment for at least 3 months.
* Concentrations of 25-oh vitamin D <20 ng / mL
* Corrected calcium <10.5 mg / dL
* Serum phosphorus <7.0 mg / dL
* Intact parathyroid hormone > 50 pg / mL and <1500 pg/mL

Exclusion Criteria:

* Active participation in another protocol.
* Vitamin D deficiency due to a hereditary disease or liver disease.
* Use of cholecalciferol ≥ 2000 IU per day within 6 months prior
* New prescription of calcitriol or paricalcitol at any dose within three months prior to the intervention (The subjects may be taking calcitriol or paricalcitol only if these drugs are taken at least three months before and no substantial changes in dosage have been made).
* Use of bisphosphonates.
* Treatment with anticonvulsants or other drugs that affect the metabolism of vitamin D.
* Pregnancy and lactation.
* Active cancer or other active inflammatory disease.
* HIV or AIDS

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-10 (Actual); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Relative reduction in serum osteoprotegerin (OPG) levels assessed by ELISA (in pg/mL) between study inclusion, and the 16-week intervention period. | 16 weeks
  The concentrations of OPG will be assessed using ELISA (Austin, Texas, USA) at inclusion and after 16 weeks of treatment with cholecalciferol or placebo.Minimum detectable concentrations for OPG are 1.9 pg/mL; intra and inter-assay coefficients of variability are 5% and 11% for OPG.

SECONDARY OUTCOMES:
Relative reduction in circulating intact fibroblast growth factor 23 (FGF23) levels (in pg/mL) | 16 weeks
  The concentrations of intact FGF-23 will be assessed using ELISA (Austin, Texas, USA)
Relative reduction in circulating osteopontin (OPN) levels (in pg/mL) | 16 weeks
  The concentrations of OPN will be assessed using ELISA (Austin, Texas, USA)
Relative reduction in circulating osteocalcin (OCN) levels (in pg/mL) | 16 weeks
  The concentrations of OCN will be assessed using ELISA ( Austin, Texas, USA)
Relative reduction in intima-media thickness measurements in the carotid artery. Ultrasound examination will be performed at study inclusion, at 16 weeks after inclusion, and up to 52 weeks post inclusion. | 52 weeks
  Ultrasound examination will be performed with the use of an 8-megahertz annular array ultrasound imaging system by a single trained sonographer. With this technique, 2 parallel echogenic lines separated by an anechoic space can be visualized at levels of the artery wall. The distance between the 2 lines gives a reliable index of the thickness of the intimal-medial complex. Subjects will be examined in the supine position. Ultrasound scans of the right and left last distal centimeter of common carotid arteries and bifurcation and of the first proximal centimeter of internal carotid arteries in 3 different projections (anterior, lateral, and posterior) will be performed. All measurements will be made at the time of scanning on unfrozen images of longitudinal scans by using the machine's electronic caliper.
Number of participants with courses of corrected calcium (>10.5 mg/dL) and phosphorus (>7 mg/dL) levels | 16 weeks
  During follow-up, all participants will be interviewed. All participants will be interviewed and a blood sample will be taken every 4-6 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Correa-Rotter, MD, Study Director — Head Dept Nephrology and Mineral Metabolism National Medical Science and Nutrition Institute Salvador Zubiran MEXICO
Locations (1):
- National Medical Science and Nutrition Institute Salvador Zubiran MEXICO, Mexico City, Mexico City, Mexico

REFERENCES:
- [Result] Ramirez-Sandoval JC, Casanova I, Villar A, Gomez FE, Cruz C, Correa-Rotter R. Biomarkers Associated with Vascular Calcification in Peritoneal Dialysis. Perit Dial Int. 2016 May-Jun;36(3):262-8. doi: 10.3747/pdi.2014.00250. Epub 2015 Aug 20. PMID 26293840
- [Result] Ammirati AL, Dalboni MA, Cendoroglo M, Draibe SA, Santos RD, Miname M, Canziani ME. The progression and impact of vascular calcification in peritoneal dialysis patients. Perit Dial Int. 2007 May-Jun;27(3):340-6. PMID 17468488
- [Result] Bhan I, Dobens D, Tamez H, Deferio JJ, Li YC, Warren HS, Ankers E, Wenger J, Tucker JK, Trottier C, Pathan F, Kalim S, Nigwekar SU, Thadhani R. Nutritional vitamin D supplementation in dialysis: a randomized trial. Clin J Am Soc Nephrol. 2015 Apr 7;10(4):611-9. doi: 10.2215/CJN.06910714. Epub 2015 Mar 13. PMID 25770176
- [Result] Van Campenhout A, Golledge J. Osteoprotegerin, vascular calcification and atherosclerosis. Atherosclerosis. 2009 Jun;204(2):321-9. doi: 10.1016/j.atherosclerosis.2008.09.033. Epub 2008 Oct 9. PMID 19007931
- [Result] Janda K, Krzanowski M, Chowaniec E, Kusnierz-Cabala B, Dumnicka P, Krasniak A, Podolec P, Sulowicz W. Osteoprotegerin as a marker of cardiovascular risk in patients on peritoneal dialysis. Pol Arch Med Wewn. 2013;123(4):149-55. doi: 10.20452/pamw.1678. Epub 2013 Mar 26. PMID 23535831